CLINICAL TRIAL: NCT02811042
Title: Laryngeal Mask Ambu AuraOnce Versus Laryngeal Mask Ambu AuraGain in Non-paralysed, Anesthetized Children: A Randomized, Crossover Study Assessing Oropharyngeal Leak Pressure and Fiberoptic Position
Brief Title: Ambu AuraOnce Versus Ambu AuraGain LM in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Schulthess Klinik (Other)
Collaborators: University of Salzburg (Other)
Responsible Party: Principal Investigator, ChristianKeller, PD Dr. med. M.Sc., Schulthess Klinik
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Schulthess_Anä_7
Record Dates: First submitted 2016-06-14; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Airway Management

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oropharyngeal leak pressure (Active Comparator): Ambu AuraOnce
  Interventions: Device: Ambu AuraOnce
- Fiberoptic position (Experimental): Ambu AuraGain
  Interventions: Device: Ambu AuraGain

INTERVENTIONS:
Device: Ambu AuraOnce — Oropharyngeal leak pressure was determined by closing the expiratory valve of the anaesthesia breathing system and a fixed gas flow of 3 l minute-1. The airway pressure at which an equilibrium was reached was noted (maximum allowed 40 cm H2O).
  Arms: Oropharyngeal leak pressure
Device: Ambu AuraGain — The airway tube view was scored using an established scoring system (4=only vocal cords visible; 3=vocal cords plus posterior epiglottis; 2=vocal cords plus anterior epiglottis; 1=vocal cords not seen)
  Arms: Fiberoptic position

SUMMARY:
The investigators test the hypothesis that oropharyngeal leak pressure and fiberoptic position differ between the size 2 LM Ambu AuraOnce and the LM Ambu AuraGain in non-paralyzed anaesthetized pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* age 1 - 16 years
* minor surgery
* extraglottic airway device

Exclusion Criteria:

* age (<12 months, >16 years)
* weight (<12 kg, >50 kg)
* a known difficult airway
* risk of aspiration

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
oropharyngeal leak pressure | 5 min

SECONDARY OUTCOMES:
fiberoptic position | 5 min

CONTACTS AND LOCATIONS:
Locations (2):
- Zentralkrankenhaus Bozen, Bolzano, Italy
- Christian Keller MD, M.Sc., Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stogermuller B, Ofner S, Ziegler B, Keller C, Moser B, Gasteiger L. Ambu(R) Aura Gain versus Ambu(R) Aura Once in children: a randomized, crossover study assessing oropharyngeal leak pressure and fibreoptic position. Can J Anaesth. 2019 Jan;66(1):57-62. doi: 10.1007/s12630-018-1235-7. Epub 2018 Oct 12. PMID 30315506